CLINICAL TRIAL: NCT04633551
Title: Supplements to Improve Vascular Inflammation After an Adverse Pregnancy Outcome
Brief Title: Vascular Inflammation and Anti-inflammatory Supplements After Adverse Pregnancy Outcomes
Acronym: VIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Abbi Danielle Lane-Cordova, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10010335
Record Dates: First submitted 2020-11-06; First posted 2020-11-18 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Pre-Eclampsia; Pre-Term; Intrauterine Growth Restriction; Hypertension in Pregnancy
Keywords: adverse pregnancy outcome; inflammation; vascular health
MeSH Terms: conditions — Pre-Eclampsia; Premature Birth; Fetal Growth Retardation; Hypertension, Pregnancy-Induced; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in this arm will receive a commercially available anti-inflammatory supplement.
  Interventions: Dietary Supplement: Anti-inflammatory supplement
- Control (No Intervention): Participants in this arm will not receive a commercially available anti-inflammatory supplement.

INTERVENTIONS:
Dietary Supplement: Anti-inflammatory supplement — commercially available combination of curcumin, quercitin, resveratrol, and green tea
  Arms: Intervention

SUMMARY:
Women who had an adverse pregnancy outcome (APO), such as preeclampsia, preterm birth, or gestational diabetes, have a higher risk for heart disease. Some of the extra risk for heart disease after APOs is thought to be caused by inflammation. Investigators will randomize women who had an APO in the past 3 years to receive an anti-inflammatory supplement or serve as a time control. Investigators will compare blood pressure, arterial stiffness, blood vessel reactivity, and blood markers of inflammation between women who did and did not receive the supplement. Investigators will determine women's attitudes about taking a dietary supplement and measure whether the participants who receive the supplement take all or most of the doses.

DETAILED DESCRIPTION:
Research Design. Investigators will invite 56 women with an APO within the past 3 yrs to participate. Women will be randomly assigned to the 4-wk intervention group (n=28) or a standard care group (n=28) using a computerized random number generator, stratified by race. Assuming up to 25% with poor adherence, Investigators expect that 42 women (21 each arm) will complete the study. No data exist related to effects of supplementation on vascular function in our population, we assumed a medium effect size, i.e. Cohen's d~0.50 and accepting a β=0.80, to generate sample sizes. Generation of effect sizes is a key outcome of this study. Investigators will conduct a vascular assessment and blood draw at two visits: before the intervention begins and within 3 days of completing the intervention. Investigators will conduct visits during the early follicular phase of menstrual cycle to account for fluctuating hormones. Vascular testing will be performed in the supine position and ≥4 hours after a light meal. Surveys for Aim 2 will be completed within the first 2 weeks of study enrollment, and interviews for Aim 2 will be conducted at the end of Visit 2.

Anti-inflammatory supplementation intervention. Participants randomized to the supplementation intervention will receive a commercially available supplement (100 mg curcumin phytosome, 100 mg quercetin phytosome, 100 mg green tea phytosome, 100 mg trans-resveratrol, 100 mg trans-pterostilbene). Participants will be asked to take 2 doses/day (1g total). Participants randomized to supplementation will receive a daily email reminding them to take the supplement. Covariates. Medical history, age, and sociodemographics will be obtained via self-report. Investigators will use validated surveys to determine physical activity, sedentary behavior, and smoking history. Height and weight will be measured.

Acceptability of Dietary Supplementation. Investigators will administer surveys to all participants to understand their perceptions of dietary supplementation, including potential benefits and consequences associated with supplementation. Investigators will determine willingness to use supplements, barriers to supplementation, and who, i.e., physician or partner, influences their decision to use dietary supplements.

Adherence and Barriers to Adherence. Investigators will count pills to determine adherence to supplementation regime. Investigators will assess each intervention participant's perceptions of supplementation with a brief interview at the final visit. Interviews will capture participant's perceptions of the role of supplementation for CVD prevention, and any side effects of supplementation. Investigators will ask participants to recommend ways to encourage participation and ask questions regarding their perceptions of the incentive structure and contact with the study team. Investigators will contact participants who drop out of the study to identify reasons for drop out.

ELIGIBILITY:
Inclusion Criteria:

* Had a singleton pregnancy in the past 3 years that lasted 20 weeks or more
* Most recent pregnancy was complicated by an APO

Exclusion Criteria:

* currently pregnant or breastfeeding,
* current smoking,
* active cancer,
* regular use of NSAIDs, steroidal medications, statins, or other anti-inflammatory supplements,
* HIV/AIDS,
* uncontrolled high blood pressure ( >160/>110 mmHg),
* unwilling or unable to use a dietary supplement,
* known sensitivity to resveratrol, curcumin, green tea, or quercetin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbi Lane-Cordova, PhD, Principal Investigator — University of South Carolina
Locations (1):
- Public Health Research Center, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
We will disseminate results at conferences and in medical journals. We are open to sharing limited datasets upon request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Upon completion of the study
Access Criteria: Contact the PI:
  Abbi Lane-Cordova lanecord@mailbox.sc.edu 803-777-7568

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 6 | 3
Completed | 5 | 3
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: There were 6 participants enrolled in the Intervention. One participant was lost to follow up and did not complete Visit 2. we analyzed data for those who completed Visit 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (6) | 30 (6) | 32 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 2 | 1 | 3
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 8
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 118 (22) | 119 (15) | 118 (18)
Arterial stiffness [Mean (Standard Deviation); unit: m/s] | 6.4 (0.5) | 8.3 (2.7) | 7.3 (1.9)
Augmentation index [Mean (Standard Deviation); unit: percentage] — Augmentation index is a measure of arterial wave reflection intensity. It is related to the heart's workload.
  percentage | 24 (6) | 25 (5) | 24 (5)
Central systolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 108 (15) | 110 (13) | 109 (14)
Reactive hyperemia [Mean (Standard Deviation); unit: ml/100 mg tissue/min] | 7.7 (3.3) | 13.2 (12.5) | 9.7 (7.7)
Inflammatory biomarker IL-6 [Mean (Standard Deviation); unit: pg/dl] — Population: We did not perform blood draws successfully on all participants.
  pg/dl
    number analyzed (Participants) | 4 | 1 | 5
    (all) | NA (NA) — Mean values for the biomarker were below detection. | NA (NA) — Mean values for the biomarker were below detection. | NA (NA) — Mean values for the biomarker were below detection.

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure (mmHg)
Description: Investigators will measure blood pressure in the arm and use applanation tonometry to estimate aortic blood pressure
Time Frame: 1 month
Population: Participants who completed Visit 2.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
mmHg | 122 (9) | 116 (9)

2. Primary Outcome: Arterial Stiffness (m/s)
Description: Arterial stiffness will be measured with pulse wave velocity using applanation tonometry and heart rate
Time Frame: 1 month
Population: Only participants who completed Visit 2.
Measure: Mean (Standard Error); unit: m/s
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
m/s | 6.2 (0.7) | 7.8 (1.2)

3. Primary Outcome: Augmentation Index (%)
Description: Applanation tonometry will be used to describe systolic blood pressure augmentation, a measure of arterial wave reflection intensity.
Time Frame: 1 month
Measure: Mean (Standard Error); unit: percentage
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
percentage | 23 (3) | 22 (4)

4. Primary Outcome: Endothelial Function (Reactive Hyperemia)
Description: Venous occlusion plethysmography will be used to mease the change in forearm blood flow after a 5-min occlusion
Time Frame: 1 month
Measure: Mean (Standard Error); unit: ml/100 mg tissue/min
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 3
ml/100 mg tissue/min | 6.6 (3.4) | 7.6 (5.6)

5. Secondary Outcome: Inflammatory Vascular Biomarkers (pg/dL)
Description: concentrations of circulating adhesion molecules ICAM and VCAM
Time Frame: 1 month
Population: Unable to perform blood draws on all participants.
Measure: Mean (Standard Deviation); unit: pg/dl
Arm/Group | Intervention | Control
Number analyzed (Participants) | 4 | 1
pg/dl | NA (NA) — Undetected values | NA (NA) — Undetected values

6. Secondary Outcome: Acceptability of Intervention (Likert Scales From 1-5; Not Likely at All to Extremely Likely and Free Text Fields)
Description: Surveys regarding opinion and likelihood of taking supplements. Here we report the number of participants who thought supplements were somewhat or extremely useful (Likert score of 4-5) for improving health.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 6 | 3
Participants | 6 | 3

7. Secondary Outcome: Perception of Intervention (15-20 Minute Interview)
Description: Interviews will be used to determine barriers and facilitators of adherence. We report number of participants who were happy with contact with study team for adherence reminders.
Time Frame: 1 month
Population: Only Intervention group participants who completed Visit 2 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 5 | 0
Participants | 5 |

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3

LIMITATIONS AND CAVEATS:
We began the study during the peak of the covid pandemic, and research capacity was limited. Recruitment was low. Target numbers were not reached.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-13): https://cdn.clinicaltrials.gov/large-docs/51/NCT04633551/Prot_SAP_000.pdf